CLINICAL TRIAL: NCT01555853
Title: A Phase I/II Institutional Study of Abraxane in Recurrent and Refractory Lymphoma
Brief Title: Phase I/II Study of Abraxane in Recurrent and Refractory Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: completed accrual to phase I but drug did not show activity, so halted before initiation of phase II
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201204071
Record Dates: First submitted 2012-03-13; First posted 2012-03-16 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin Disease
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase I-Dose Level 0 (Experimental): Abraxane 100 mg/m2 IV on Days 1, 8, and 15 of each 28 day cycle for a maximum of 6 cycles.
  Interventions: Drug: Abraxane
- Phase I-Dose Level 1 (Experimental): Abraxane 125 mg/m2 IV on Days 1, 8, and 15 of each 28 day cycle for a maximum of 6 cycles.
  Interventions: Drug: Abraxane
- Phase I-Dose Level 2 (Experimental): Abraxane 150 mg/m2 IV on Days 1, 8, and 15 of each 28 day cycle for a maximum of 6 cycles.
  Interventions: Drug: Abraxane
- Phase II (Experimental): Abraxane (dose to be determined in Phase I) IV on Days 1, 8, and 15 of each 28 day cycle for a maximum of 6 cycles.
  Interventions: Drug: Abraxane

INTERVENTIONS:
Drug: Abraxane
  Other Names: ABI-007

SUMMARY:
This phase I/II trial studies the side effects, maximum tolerated dose, and effectiveness of paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel) in treating patients with recurrent or refractory Hodgkin or B-cell non-Hodgkin lymphoma. More effective and well tolerated therapies are needed to treat patients with relapsed and refractory lymphomas. Nab-paclitaxel combines a chemotherapeutic agent with a protein which may increase the anticancer drug concentration in the tumor while reducing toxic effects in normal tissue and may be an effective treatment for lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed B-cell non-Hodgkin lymphoma or classical Hodgkin lymphoma:

  * Diffuse large B-cell lymphoma (including transformed large cell lymphoma and primary mediastinal B cell lymphoma)
  * Mantle cell lymphoma
  * Burkitt's lymphoma
  * Follicular lymphoma
  * Small lymphocytic lymphoma
  * Marginal zone lymphoma
  * Lymphoplasmacytic lymphoma
  * Classical Hodgkin lymphoma (including nodular sclerosis, mixed cellularity, lymphocyte rich, and lymphocyte deplete)
* Patient must have measurable disease, defined as the presence of ≥ 1 lymph node or tumor mass measuring ≥ 1 cm in a single dimension as assessed by CT or MRI.
* Patient must have had prior treatment with ≥ 2 chemotherapy or chemo-immunotherapy regimens. Prior autologous stem cell transplant is allowed, and prior allogeneic stem cell transplant is allowed as long as the patient has recovered from acute toxicities and is off immunosuppression without evidence of graft versus host disease (GVHD).
* Patient must be ≥ 18 years of age.
* Patient must have an ECOG performance status ≤ 2.
* Patient must have adequate bone marrow reserve at the time of therapy initiation, defined as ANC ≥ 1.0 x 109/L and platelets ≥ 50 x 109/L.
* Patient must have adequate hepatic function, defined as total bilirubin ≤ 1.5 x ULN and AST/ALT ≤ 3 x ULN.
* Patient must have adequate renal function, defined as serum creatinine ≤ 2.0 x ULN.
* Patient must have recovered from any acute toxicities associated with prior therapy to ≤ grade 1.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patient (or legally authorized representative, if applicable) must be able to understand and willing to sign an IRB approved written informed consent document.
* Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patient must not have nodular lymphocyte predominant Hodgkin lymphoma subtype.
* Patient must not have a history of a non-lymphoma malignancy except for the following: adequately treated localized basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, superficial bladder cancer, localized prostate cancer, any adequately treated stage I or stage II cancer currently in complete remission, or any other cancer in complete remission for at least 5 years.
* Patient must not be receiving any other investigational agents, and must not have taken any other investigational agents within ≤ 3 weeks of study entry chemotherapy, immunotherapy, radiotherapy, and/or investigational agents while on study.
* Patients with Hodgkin's lymphoma must not otherwise be eligible for treatment with brentuximab vedotin.
* Patient must not have central nervous system or leptomeningeal lymphoma.
* Patient must not have with history of allergic reactions attributed to compounds of similar chemical or biologic composition to Abraxane.
* Patient must not have any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not be pregnant and/or breastfeeding.
* Patient must not be known to be HIV-positive.
* Patient must not have any pre-existing peripheral neuropathy > grade 1.
* Patient must not have received any chemotherapy, immunotherapy, and/or investigational agents and/or radiotherapy < 3 weeks prior to starting study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose (MTD) of Abraxane in patients with recurrent or refractory lymphoma | 28 days (completion of cycle 1) for all patients in Phase I portion
  Graded and described using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4.
Phase I: Dose-limiting toxicities (DLTs) of Abraxane in patients with recurrent or refractory lymphoma | 28 days (completion of cycle 1)
  Graded and described using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4
Phase II: Overall response rate (CR + PR) | 24 weeks (end of study)

SECONDARY OUTCOMES:
Phase I: Toxicity associated with Abraxane | 28 weeks (30 days after completion of study treatment)
Phase II: Time to progression. | 24 weeks (end of study)
  Response and progression will be recorded with each imaging evaluation according to the 2007 revised response criteria for malignant lymphoma by Cheson BD, Pfistner B, Juweid ME, et al. Revised response criteria for malignant lymphoma. J Clin Oncol 2007;25:579-86.
Phase II: Duration of remission | 24 weeks (end of study)
Phase II: Overall survival. | 3 years
Phase II: Clinical benefit (CR + PR + SD) | 24 weeks (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bartlett, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - St. Louis University School of Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu